CLINICAL TRIAL: NCT07029581
Title: A Double-Blind, Placebo-Controlled, Phase 2, Efficacy and Safety Study of ACP-204 in Adults With Lewy Body Dementia Psychosis (LBDP)
Brief Title: Phase 2, Efficacy and Safety Study of ACP-204 in Lewy Body Dementia Psychosis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: ACADIA Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ACP-204-012; 2025-521710-25-00 (EU CTIS Number)
Record Dates: First submitted 2025-06-12; First posted 2025-06-19 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2025-09

CONDITIONS: Lewy Body Dementia Psychosis

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized to one of 3 parallel arms i.e. ACP-204 at one of 2 dose levels (30 or 60 mg) or placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- ACP-204 30 mg (Experimental): ACP-204 dose of 30 mg once daily
  Interventions: Drug: ACP-204
- ACP-204 60 mg (Experimental): ACP-204 dose of 60 mg once daily
  Interventions: Drug: ACP-204
- Placebo (Placebo Comparator): Placebo once daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ACP-204 — Provided as 1 capsule, to be taken orally once daily
  Arms: ACP-204 30 mg; ACP-204 60 mg
Drug: Placebo — Provided as 1 capsule, to be taken orally once daily
  Arms: Placebo

SUMMARY:
Multicenter, randomized, 6-week, double-blind, placebo-controlled, parallel-group, Phase 2 study in subjects with LBDP.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥55 years to <85 years of age at the Screening visit living in the community or, if permitted by local regulations, in an institutionalized setting
* Can provide written informed consent. If the subject is deemed not competent to provide informed consent, the following requirements for consent must be met:

  1. The subject's LAR must provide written informed consent.
  2. The subject must provide written (if capable) informed assent per local regulations.
* Meets either the clinical criteria for Parkinson's disease with dementia as defined by the Movement Disorder Society's Task Force or the revised clinical criteria for probable dementia with Lewy bodies (DLB) by consensus criteria (Fourth consensus report of the DLB Consortium).
* Meets the revised criteria for psychosis in major or mild neurocognitive disorder established by the International Psychogeriatrics Association

Exclusion Criteria:

* Is in hospice, is receiving end-of-life palliative care, or is bedridden
* Has psychotic symptoms that are primarily attributable to delirium, substance abuse, or a medical or psychiatric condition (e.g. schizophrenia, bipolar disorder, delusional disorder) other than dementia
* Is actively suicidal at Visit 1 (Screening) or Visit 2 (Baseline)
* Has a history or current evidence of a serious and/or significant unstable cardiovascular, respiratory, endocrine, gastrointestinal, renal, hepatic, hematologic, immunologic, genitourinary, psychiatric or neurologic (including stroke, chronic seizures, or clinically significant head injury) abnormality or disease or other medical disorder, including cancer or malignancies that could interfere with subject's ability to complete the study or comply with study procedures
* Has other clinically significant CNS abnormalities that are most likely contributing to the dementia or findings on MRI or CT

Ages: 55 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-08-06 (Actual); Primary Completion 2028-02 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in SAPS-LBDP total score at Week 6 | 6 weeks
  Change from Baseline in Scale for the Assessment of Positive Symptoms- Lewy Body Dementia Psychosis (SAPS-LBDP) total score at Week 6

CONTACTS AND LOCATIONS:
Locations (37):
- United States (21):
  - ATP Clinical Research Inc., Irvine, California
  - Humanity Clinical Research, Corp, Aventura, Florida
  - Parkinson's Disease and Movement Disorders Center of Boca Raton, Boca Raton, Florida
  - K2 Medical Research Winter Garden LLC, Clermont, Florida
  - K2 Summit Research, Lady Lake, Florida
  - Neurology Associates, P. A., Maitland, Florida
  - Homestead Associates in Research Inc, Miami, Florida
  - Premier Clinical Research Institute, Inc., Miami, Florida
  - Advanced Clinical Research Network, Corp, Miami, Florida
  - MediClear Medical & Research Center, Inc., Miami, Florida
  - Health Synergy Clinical Research, LLC, West Palm Beach, Florida
  - Hawaii Pacific Neuroscience, Honolulu, Hawaii
  - University of Kansas Medical Center Research Institute Inc., Kansas City, Kansas
  - Parkinson's Disease and Movement Disorders Center of Boca Raton d/b/a Parkinson's Research Center of America-Long Island, Commack, New York
  - The Ohio State University, Energy Advancement and Innovation Center, Columbus, Ohio
  - The Movement Disorder Clinic of Oklahoma, Tulsa, Oklahoma
  - Abington Neurological Associates, LTD, Abington, Pennsylvania
  - Horizon Clinical Research Group, Cypress, Texas
  - The University of Texas Health Science Center San Antonio, San Antonio, Texas
  - R and H Clinical Research, Stafford, Texas
  - Virginia Commonwealth University (a public institution of higher education), Richmond, Virginia
- Bulgaria (5):
  - Ambulatory for Individual Practice for Specialized Medical Care in Psychiatry - Dr Ivo Natsov, Cherven Bryag
  - UMHAT Sv Georgi EAD, Plovdiv
  - Medical Center SV.Naum, Sofia
  - Medical Center Detsko Zdrave Branch Maestro Kanev, Sofia
  - DCC Mladost M- Varna, OOD, Varna
- Czechia (5):
  - Fakultni nemocnice u sv. Anny v Brne, Brno
  - NEUROHK s.r.o. Poliklinika Chocen a.s., Choceň
  - Vseobecna fakultni nemocnice v Praze, Prague
  - Neuropsychiatrie s.r.o., Prague
  - Vestra Clinics s.r.o, Rychnov nad Kněžnou
- France (4):
  - Hopital Neurologique Bron, Bron
  - Hopital BROCA, Paris
  - CHU Strasbourg-Hopital Hautepierre, Strasbourg
  - CHRU de Tours- Hopital Bretonneau, Tours
- Serbia (2):
  - Institute of Mental Health, Belgrade
  - University Clinical Center of Serbia, Belgrade

IPD SHARING:
Plan to Share IPD: No